CLINICAL TRIAL: NCT06895603
Title: The HIgh-fidelity Hydraulic couPling Upper-arm Cuff Assessment of Limits, Safety, and Effectiveness (HIPULSE) Trial (Cardiac Output Study)
Acronym: CO
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: HIPULSE-CO_PAC_2021_11366
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: ICU; Surgical Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All patients being monitored with a pulmonary artery catheter: Up to 75 intensive care unit patients being monitored with a pulmonary artery catheter (approximately 20 patients from at least 2 sites during the roll-in phase and approximately 55 patients during the pivotal phase) will be enrolled over an estimated 8 months accrual and follow-up evaluation period. There will be no randomization in this study.
  Interventions: Device: Philips Advanced Monitoring Cuff (AMC)

INTERVENTIONS:
Device: Philips Advanced Monitoring Cuff (AMC) — The Philips AMC is a Class II (USA) and Class IIb (EU) medical device that is a non-invasive, semirigid disposable upper arm cuff with an integrated pneumatic actuator enabling hydraulic coupling of tissue pressure waveforms from the upper arm tissue.

SUMMARY:
The purpose of this study is to compare cardiac output (CO), fluid responsiveness, and related measurements between the Philips AMC and PAC (Swan-Ganz) in ICU or surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Indication for PAC (Swan-Ganz)
* Indication for radial arterial line
* Subject or legal authorized representative is able to understand and speak the local language (also Spanish is also accepted for US sites) to provide voluntary written informed consent prior to study procedures

Exclusion Criteria:

* Emergency surgery
* ICU or surgical positioning where both arms are tucked
* Inability to place the Philips AMC appropriately due to subject anatomy or condition
* Known pregnancy or lactating women (self-report)
* Patients treated with an intra-aortic balloon pump
* Measurements taken in the lateral position
* Currently participating in an investigational drug or another device study that clinically interferes with the study endpoints
* Upper arm circumference < 19 cm or > 43 cm
* BMI > 45
* At the PI's discretion, subject does not qualify to participate in the study for any reasons that are not mentioned above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 75 ICU patients being monitored with a PAC and radial arterial line will be enrolled over approximately 8 months accrual and follow-up evaluation period
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoints | Approximately 8 months for accrual and follow-up
  The comparison of cardiac output between the Philips AMC and PAC

CONTACTS AND LOCATIONS:
Locations (2):
- UVA Health, Charlottesville, Virginia, United States
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No